CLINICAL TRIAL: NCT04449120
Title: HOME COOKING: Health Empowerment Strategy in People With Type II Diabetes Mellitus (SUKALMENA)
Brief Title: HOME COOKING: Health Empowerment Strategy in People With Type II Diabetes Mellitus
Acronym: SUKALMENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Culinary Center Fundazioa (Other)
Collaborators: University of Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04.0006.19
Record Dates: First submitted 2020-06-19; First posted 2020-06-26 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Mediterranean diet; Culinary intervention; Cooking classes; Home cooking
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study uses a randomized controlled trial design with one-month intervention program and three months of follow-up in order to test the effects of a culinary intervention program to improve cooking and healthy eating behaviour in type 2 diabetic patients.
  The culinary intervention program will be given over a one-month period, one day a week for four weeks. Participants in the control group (CG) will receive dietary training based on Mediterranean diet at the baseline visit and a leaflet explaining this dietary pattern. The participants assigned to the culinary intervention program will receive the same nutritional recommendations and four online cooking classes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional education group (NEG) (Active Comparator): Participants in the nutritional education group will be given a leaflet with written nutrition educational information to follow a Mediterranean diet. Participants will be encouraged to adhere to this diet for one-month. Three visits will be scheduled for participants assigned to this group:
  (1) before randomization (T1); (2) after randomization and before the program´s beginning (T2); and (3) after three months of follow-up period. In all time-points, questionnaires will be registered and at T2 and T3 blood samples will be collected. Volunteers will be contacted by phone after 1 month and 6 months of the end of the intervention to collect information about food and culinary habits.
  Interventions: Behavioral: Mediterranean diet-based nutritional education intervention
- Culinary intervention group (CIG) (Experimental): Participants assigned to the culinary intervention group received the written nutrition educational information as well as four online cooking classes (one cooking class per week) during the one-month intervention period. Three visits will be scheduled for participants assigned to this group:
  (1) before randomization (T1); (2) after randomization and before the program´s beginning (T2); and (3) after three months of follow-up period. In all time-points, questionnaires will be registered and at T2 and T3 blood samples will be collected.
  Participants will attend 4 culinary workshops between visit 2 and 3. Volunteers will be contacted by phone after 1 month and 6 months of the end of the intervention to collect information about food and culinary habits.
  Interventions: Behavioral: Mediterranean diet-based culinary intervention

INTERVENTIONS:
Behavioral: Mediterranean diet-based culinary intervention — The culinary intervention was developed integrating four culinary workshops that were given every week, once per week, during one-month intervention. The duration of each culinary workshop was 3,5 h, thus, the program provided a total of 14h of practice in cooking activities. The courses took place in a well-equipped kitchen from the Basque Culinary Center. Each culinary workshop was divided in two differentiated parts in order to work on the specific objectives established for each day. All cooking classes began with a theoretical introductory part that aimed to explain the main take-home messages from the workshop. Subsequently, every class was characterized by a hands-on part that included the demonstration and practical preparation of different elaborations based on the use specific cooking techniques and healthy ingredients. At the end of the session, participants were encouraged to taste the prepared meals, to share their preferences and their view about the cooking experience.
  Arms: Culinary intervention group (CIG)
Behavioral: Mediterranean diet-based nutritional education intervention — The patients in the nutritional intervention group will receive dietary advice on how to follow a Mediterranean diet. The dietary recommendations will be given at the beginning of the study by nutritionists using comprehensive written material.
  Arms: Nutritional education group (NEG)

SUMMARY:
Currently, one of the health challenges in the field of public health is to improve the quality of life of people with metabolic diseases, using new strategies that allow to promote healthy eating habits.

Within the new strategies that may encourage population improving eating habits, "HOMECOOKING" is proposed as a transforming tool for health, involving culinary skills and knowledge in nutrition. It is suggested as a new paradigm in nutritional education.

This project will cover the "HOMECOOKING: cooking and eating at home", as an innovative strategy, aiming to improve the quality of the diet of people with type II diabetes mellitus through an intervention based on cooking workshops. At these sessions, participants will learn easy cooking techniques and tools, in order to acquire culinary competences and to be empowered to prepare healthy dishes.

The effect of this intervention programme on the health of the participants will be evaluated through the measurement of biochemical parameters related to the disease (glycosylated haemoglobin, insulin, glucose, among others). In addition, specific compounds known as advanced glycation end products (AGEs) will be measured. The formation of these compounds is associated with the type of food consumed and the culinary techniques that are applied.

DETAILED DESCRIPTION:
One of the main factors influencing health is nutrition. Therefore, lifestyle and more specifically healthy eating habits, are key elements for the promotion of healthy lifestyle in society. Eating habits are defined as the more or less conscious, collective and repetitive behaviour that leads people to select, consume and use a certain foods or diet, in response to social and/or cultural influences. The acquisition of eating habits occurs since childhood. For this reason, an education in food and gastronomy is necessary to promote healthy eating habits in society. Education programmes so far have focused on nutrition education, i.e. on transferring theoretical knowledge about nutrition. However, currently, it is known that traditional knowledge about nutrition is not sufficient and it is necessary to go deeper into the factors that determine what people eat, and how people eat.

The studies related to the sensory perception of food and the relationship that this perception has with the choice of food, seek to decipher the keys that make different individuals to have certain eating habits based on: personal tastes, the influence of culture, the emotions that make them feel, learning, and so on. Nutritional recommendations will always be simpler to follow when, implicit in them, the tastes and food choices of each individual are found.

From a holistic perspective, individuals should be considered as a human being within a social, cultural and technological environment. In this sense, gastronomy is defined as "the reasoned knowledge of what people eat and how people eat. It is an interdisciplinary area of knowledge that studies and generates physical-chemical, cultural and socioeconomic processes where human beings cultivate, process, distribute and consume good foods and beverages that affect their physical, mental and social well-being". Gastronomy is a vehicle capable of creating social trends and the convergence of this discipline together with nutritional education can be a more effective tool to disseminate messages about what is considered a healthy diet, how to eat a healthy diet, as well as to transfer cooking skills that allow the population to acquire and sustain these eating habits at home.

Briefly, gastronomy plays a fundamental role in covering the nutritional needs of the general population, and at the same time, it satisfies their expectations of flavour. Therefore, gastronomy is considered a decisive channel to favour education of taste, a better nutrition and, in general, for health promotion.

The effect of nutrition on health is not homogeneous in the population. On the one hand, factors such as the type of food and the culinary techniques used have an influence. On the other hand, individual characteristics such as lifestyle, genetic background and wellbeing must be taken into account. In this context, Personalized and Precision Gastronomy based on individuals' eating habits, genetic profile, intestinal microbiota profile, metabolome, epigenome, tastes and preferences, and so on, in order to develop strategies that favour a healthy and tailor-made diets for each individual.

Type 2 diabetes mellitus (T2DM) is one of the most prevalent metabolic diseases worldwide. In the Basque Country, it is estimated that the disease affects 10% of the population. People with diabetes have a high risk of suffering complications related to this illness. In addition, people with T2DM are more prone to develop other diseases such as cardiovascular diseases as well as premature mortality. For this reason, it is necessary to prevent the disease and to try to reduce the risk of developing complications in people who have already been diagnosed with T2DM.

The current increase in DMT2 is associated with an increase in obesity. This multifactorial disease, in turn, has been related to unhealthy lifestyles. Moreover, apart from physical activity, following a healthy diet is a determining factor. Although there is increasing information on nutrition, the desired effect on the prevention of this disease is not being achieved. This may in part be due to a lack of skills to continue a healthy diet.

Attention should also being paid to individual factors that may influence in specific nutritional needs of T2DM. In this sense, personalised gastronomy can facilitate the empowerment of people with diabetes providing them with culinary techniques and skills that allow patients to follow a healthy diet adapted to the conditions of this disease and to personal needs and preferences.

In this context, the HOME COOKING project seeks to carry out a one-month culinary intervention programme with people diagnosed with T2DM, in order to analyse the health effects that the programme can produce, comparing it with the results obtained with a traditional intervention solely based on the training of theoretical recommendations about nutrition.

In conclusion, the main hypothesis of this project lies in the fact that one of the barriers for the population to acquire and maintain healthy eating habits is related, in part, to the fact that they do not have enough culinary skills (food preparation) and do not have sufficient knowledge about nutrition (knowledge about the product). Thus, bearing in mind that several studies have demonstrated the relationship between the trust (empowerment) that provides to have food preparation skills (culinary skills), and knowledge about the quality of the diet in terms of health, the present project suggests that beneficial effects on health can be obtained when nutritionists and public health professionals promote culinary intervention programmes aimed at providing theoretical and practical knowledge.

Therefore, this project is novel since it proposes a paradigm shift promoting the incorporation of culinary training as a complement to nutritional education. Likewise, the project is based on the Mediterranean diet, a diet pattern whose health benefits have been scientifically endorsed. The study is a reference project in this field and its results will be of great relevance to public health.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 Diabetes Mellitus without treatment with insulin, sulfonylureas and glinides.
* Overweight or obesity (BMI between 25 and 40 kg/m2).
* Stable treatment with oral antidiabetics, other than sulfonylureas or glinides, at least for 3 months.

Exclusion Criteria:

* Treatment with insulin, sulfonylureas or glinides
* Glycosylated hemoglobin (HbA1c) concentration greater than 10%
* Weight loss exceeding 5 kg in the past three months
* Pregnant or breastfeeding women
* Serious medical condition that impedes from conducting the dietary intervention or that limits the survival to less than one year
* Consumption of illegal drugs, chronic alcoholism or alcohol total consumption above 80 g/day
* Participation in other clinical trial with drugs or nutritional intervention during the previous year to inclusion
* Major difficulties or inconveniences in changing dietary habits and following the Mediterranean Diet (allergies, intolerances)
* Difficulties for regular home cooking and/or eating out more than 2 days per week
* Current diagnosis of an eating disorder, schizophrenia, other psychotic disorder or bipolar disorder
* Hospitalization for any mental illness in the previous year
* History of bariatric surgery or extensive bowel resection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change in fasting glycosylated hemoglobin level | Baseline; three months follow-up
  At baseline blood samples will be collected for determination of hemoglobin A1c. At 3 months of follow-up, the determination of this parameter will be repeated.
Change in fasting glucose level | Baseline; three months follow-up
  At baseline blood samples will be collected for determination of fasting glucose levels. At 3 months of follow-up, the determination of this parameter will be repeated.
Change in fasting insulin level | Baseline; three months follow-up
  At baseline blood samples will be collected for determination of fasting insulin levels. At 3 months of follow-up, the determination of this parameter will be repeated.

SECONDARY OUTCOMES:
Change in advanced glycation end products (AGEs) level | Baseline; three months follow-up
  At baseline blood samples will be collected for determination of advanced glycation end products levels. At 3 months of follow-up, this determination will be repeated.
Changes in hip circumference | Baseline; three months follow-up
  At baseline, hip circumference will be measured with a measuring. At 3 months of follow-up , the determination of this measurement will be repeated.
Changes in waist circumference | Baseline; three months follow-up
  At baseline, waist circumference will be measured with a measuring. At 3 months of follow-up , the determination of this measurement will be repeated.
Changes in body mass index (BMI) | Baseline; three months follow-up
  BMI will be calculated as body weight (kg) divided by height (m) squared at baseline and at 3 months of follow up.
Change in fat mass | Baseline; three months follow-up
  At baseline and at 3 months of follow-up, fat mass will be analyzed by bioimpedance.
Change in fat free mass | Baseline; three months follow-up
  At baseline and at 3 months of follow-up, fat free mass will be analyzed by bioimpedance.
Changes in lipid metabolism parameters | Baseline; three months follow-up
  At baseline blood samples will be collected for determination of in fasting total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides levels. At 3 months of follow-up, the determination of these parameters will be repeated.
Change in blood pressure | Baseline; three months follow-up
  At baseline systolic blood pressure and diastolic blood pressure will be reported in mmHg.
  At 3 months of follow-up, the determination of systolic and diastolic blood pressure will be repeated.
Change in plasma C-reactive protein | Baseline; three months follow-up
  At baseline blood samples will be collected for determination of C-reactive protein. At 3 months of follow-up, the determination of this parameter will be repeated.
Change in adherence to the Mediterranean Diet measured by Mediterranean Diet Adherence Screener | Baseline; one month; three months follow-up
  At baseline data about adherence to the Mediterranean Diet will be collected by a 14-point Mediterranean Diet Adherence Screener (MEDAS). At 1 and 3 months of follow-up these data will be also collected.
Change in dietary intake measured by validated Food Frequency Questionnaire (FFQ) | Baseline; three months follow-up
  At baseline data about dietary intake will be collected by using a Food Frequency Questionnaire (FFQ). At 3 months of follow-up, these data will be also collected.
Change in quality of life measured by Quality of Life Questionnaire | Baseline; three months follow-up
  At baseline and at 3 months of follow-up, data about quality of life will be measured by Quality of Life Questionnaire.
Change in physical activity level measured by the Minnesota Leisure-Time Physical Activity Questionnaire | Baseline; three months follow-up
  At baseline and at 3 months of follow-up, data about physical activity level will be collected by the Minnesota Leisure-Time Physical Activity Questionnaire
Change in culinary habits measured by Culinary Habits Frequency Questionnaire (CHFC) | Baseline; three months follow-up
  At baseline and at 3 months of follow-up, data about culinary habits will be collected by culinary habits frequency questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Usune Etxeberria, PhD, Principal Investigator — Basque Culinary Center Fundazioa
Locations (1):
- Basque Culinary Center, Donostia / San Sebastian, Guipuzcoa, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernardo GL, Jomori MM, Fernandes AC, Colussi CF, Condrasky MD, Proenca RPDC. Nutrition and Culinary in the Kitchen Program: a randomized controlled intervention to promote cooking skills and healthy eating in university students - study protocol. Nutr J. 2017 Dec 20;16(1):83. doi: 10.1186/s12937-017-0305-y. PMID 29262811
- [Background] Reicks M, Kocher M, Reeder J. Impact of Cooking and Home Food Preparation Interventions Among Adults: A Systematic Review (2011-2016). J Nutr Educ Behav. 2018 Feb;50(2):148-172.e1. doi: 10.1016/j.jneb.2017.08.004. Epub 2017 Sep 25. PMID 28958671
- [Background] Byrne C, Kurmas N, Burant CJ, Utech A, Steiber A, Julius M. Cooking Classes: A Diabetes Self-Management Support Intervention Enhancing Clinical Values. Diabetes Educ. 2017 Dec;43(6):600-607. doi: 10.1177/0145721717737741. Epub 2017 Oct 19. PMID 29047323
- [Background] Irl B H, Evert A, Fleming A, Gaudiani LM, Guggenmos KJ, Kaufer DI, McGill JB, Verderese CA, Martinez J. Culinary Medicine: Advancing a Framework for Healthier Eating to Improve Chronic Disease Management and Prevention. Clin Ther. 2019 Oct;41(10):2184-2198. doi: 10.1016/j.clinthera.2019.08.009. Epub 2019 Sep 20. PMID 31543284
- [Background] Polak R, Tirosh A, Livingston B, Pober D, Eubanks JE Jr, Silver JK, Minezaki K, Loten R, Phillips EM. Preventing Type 2 Diabetes with Home Cooking: Current Evidence and Future Potential. Curr Diab Rep. 2018 Sep 14;18(10):99. doi: 10.1007/s11892-018-1061-x. PMID 30218282